CLINICAL TRIAL: NCT05120778
Title: Effectiveness of Exercise Training on Health and Medical Costs of Metabolic Syndrome Factors in the Adult Population.
Brief Title: Exercise Training on Health and Medical Costs of Metabolic Syndrome Individuals.
Acronym: EXEisMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 8211121078-121078-57-421
Record Dates: First submitted 2021-09-27; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; exercise training; healthcare cost; high-intensity interval training; strength training
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Cluster randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional medical treatment (Experimental): Volunteers will maintain habitual medical treatment.
  Interventions: Other: conventional medical treatment
- exercise training + conventional medical treatment (Experimental): Volunteers will maintain habitual medical treatment and will participate in a 16-week exercise training based on high-intensity interval training (stationary bikes), and strength training (weight-bearing exercises).
  Interventions: Behavioral: exercise training; Other: conventional medical treatment

INTERVENTIONS:
Behavioral: exercise training — as appear in arm description.
  Arms: exercise training + conventional medical treatment
Other: conventional medical treatment — participants will maintain habitual medical treatment prescribed by primary care and specialized physicians from the public health service.

SUMMARY:
The purpose of this study is to determine if an exercise training intervention together with conventional medical treatment can decrease the annual healthcare cost in patients with metabolic syndrome.

DETAILED DESCRIPTION:
It is proposed a multicentral clinical trial with cluster randomization among research nodes located in towns of Castilla-La Mancha and Toledo neighborhoods (Spain). The aim is to compare the annual healthcare cost of patients receiving conventional medical treatment against patients receiving the same intervention plus exercise training for 16 weeks. Exercise training will be based on high-intensity interval training conducted on stationary bikes, and strength training using weight-bearing exercises. Each research node will be composed of the clinical center and the sports facilities available in the town/neighborhood. Research nodes will be randomized into two experimental interventions: i.) conventional medical treatment, and ii.) conventional medical treatment + exercise training. After verbal and written information about the study and related potential risks, all patients fulfilling inclusion criteria will be included after giving written informed consent. At baseline, and after 12 and 24 months, annual healthcare costs will be obtained from the volunteers' clinical records. In addition, at baseline, and after 4, 12, and 24 months, metabolic syndrome components prevalence, metabolic syndrome z-score, body composition, and cardiorespiratory fitness will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling criteria for metabolic syndrome diagnosis.

Exclusion Criteria:

* At baseline, engagement to an exercise training program for the last 6 months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Annual healthcare cost | Baseline, month 12 and 24
  From unified medical records, all clinical and paraclinical interventions including pharmacological treatment, diagnostic or therapeutic procedures and primary care and specialized medical consultations will be included

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Baseline, month 4,12, and 24.
  Estimation of vo2max from a graded exercise test plus a verification test
Body composition | Baseline, month 4,12, and 24.
  Measurement of the mass of man body compartments (i.e., fat mass, fat free mass, and bone mass) by dual energy x-ray absorptiometry.
Blood lipids profile | Baseline, month 4,12, and 24.
  Serum concentrations (in mg per dL) of triglycerides, total colesterol, high density lipoprotein after 8-hour fasting
Glycemia | Baseline, month 4,12, and 24.
  Serum concentrations of glycemia (in mg per dL) after 8-hour fasting
Blood pressure | Baseline, month 4,12, and 24.
  Systolic and diastolic values of blood pressure measures obtained from the brachial artery after 15 min of supine rest.
Central obesity | Baseline, month 4,12, and 24.
  Measurement of waist circumference (cm) in a horizontal plane, midway between the inferior margin of the ribs and the superior border of the iliac crest.

OTHER OUTCOMES:
Compliance to Exercise volume prescription . | Month 4
  From the exercise training sessions records (exercise time in minutes), measurement of volume prescription (Target time)
compliance to Exercise intensity prescription. | Month 4
  From the exercise training sessions records (heart rate in beats per minute), measurement of compliance to exercise intensity prescription (target HR).
Daily physical activity | Month 4,12, and 24.
  Measurement of daily steps using pedometers

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Mora-Rodriguez, PhD, Principal Investigator — University of Castilla-La Mancha

IPD SHARING:
Plan to Share IPD: No